CLINICAL TRIAL: NCT03782064
Title: A Phase II Trial of Vaccination With Dendritic Cell (DC)/Myeloma Fusions in Combination With Nivolumab in Patients With Relapsed Multiple Myeloma
Brief Title: Dendritic Cell (DC)/Myeloma Fusions in Combination With Nivolumab in Patients With Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-280
Record Dates: First submitted 2018-12-13; First posted 2018-12-20 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+DC/myeloma fusions/GM-CSF (Experimental): * Nivolumab will be given every two weeks
  * The DC/myeloma fusion vaccine/GM-CSF is administered 4 days per cycle
  Interventions: Drug: Nivolumab; Biological: DC/myeloma fusions/GM-CSF

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a monoclonal antibody. Antibodies are part of your immune system; they are a type of protein that protects your body against foreign invaders, called antigens, by grabbing hold of antigens to stop them from invading your system. Nivolumab has been shown to react against cancer cells, including MM cells.
Biological: DC/myeloma fusions/GM-CSF — The DC/MM vaccine is an investigational agent that tries to help the immune system recognize and fight against cancer cells, utilizing unique markers.

SUMMARY:
This research study is studying a cancer vaccine called Dendritic Cell/MM Fusion vaccine (DC/MM vaccine) in combination with nivolumab, as a possible treatment for multiple myeloma (MM).

The drugs involved in this study are:

* Dendritic Cell/MM Fusion vaccine (DC/MM vaccine)
* Nivolumab, an immunotherapy drug

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the DC/MM vaccine as a treatment for any disease.

The FDA has not approved nivolumab for multiple myeloma. A similar immunotherapy drug used in combination with IMiDs (drugs that regulate or modify the immune system) was associated with higher risk of death in another research trial in patients with multiple myeloma; however, nivolumab has been approved for use in several other types of cancers.

The FDA has not approved the combination of nivolumab with the DC/MM vaccine as a treatment for any disease.

In this research study, the investigators wish to determine whether nivolumab administered in combination with the DC/MM vaccine will help promote an immune response against multiple myeloma cells.

An immune response is any reaction by the immune system. It helps the body distinguish itself from substances foreign to it, such as infections and dangerous substances. Cancer cells have unique markers that distinguish them from normal cells, which can potentially serve as targets for the immune system.

The DC/MM vaccine is an investigational agent that tries to help the immune system recognize and fight against cancer cells, utilizing those unique markers. Unlike a standard vaccine that is used to prevent infections, cancer vaccines are being studied to see if they can fight cancers that are already in the body. Laboratory studies suggest that when dendritic cells (a type of immune cell that helps to tell your immune system what is good and what is bad) and tumor cells are brought together, the dendritic cells can stimulate immune responses against the tumor.

Nivolumab is a monoclonal antibody. Antibodies are part of your immune system; they are a type of protein that protects the body against foreign invaders, called antigens, by grabbing hold of antigens to stop them from invading your system. Monoclonal indicated that this antibody was made in a lab. Nivolumab has been shown to react against cancer cells, including MM cells. The investigators hope that the addition of nivolumab with the DC/MM vaccine will help the body fight MM

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Patients with relapsed multiple myeloma with prior treatment of an IMID and proteasome inhibitor.
* Age ≥18 years.
* ECOG performance status ≤2
* Patients must have > 20% plasma cells in the bone marrow aspirate differential <30 days prior to enrollment.
* ANC > 1000; Platelets > 75K without transfusional support
* Participants must have normal organ function as defined below:

  * total bilirubin ≤1.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal
  * creatinine clearance ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of DC/MM fusion and nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 5 months after completion of treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

-Participants who are receiving any other investigational agents.

3.2.2 Patients with purely non-secretory MM [absence of a monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence-Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques and the absence of involved serum free light chain >100 mg/L]. Patients with light chain MM detected in the serum by free light chain assay are eligible.

* Patients with Plasma Cell Leukemia
* Because of compromised cellular immunity, patients who have a known human immunodeficiency virus (HIV), active hepatitis C virus (HCV) or active hepatitis B virus (HBV).
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure (see Appendix H), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening will be documented by the investigator as not medically relevant.
* Active or prior documented autoimmune or inflammatory disorders including but not limited to the following:

  * GI Disorders: (including inflammatory bowel disease [e.g. ulcerative colitis, Crohn's disease], diverticulitis (with the exception of a prior episode that has resolved), celiac disease, or other serious gastrointestinal chronic conditions associated with diarrhea.
  * Systemic lupus erythematosus
* Wegener's syndrome [granulomatosis with polyangiitis]

  * Myasthenia gravis
  * Graves' disease
  * Rheumatoid arthritis
  * Hypophysitis
  * Uveitis
* The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Note: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: non-invasive cancer (such as, any in situ cancers) and basal cell or squamous cell carcinoma of the skin.
* Female patients who are pregnant (positive β-HCG) or breastfeeding
* Prior organ transplant requiring immunosuppressive therapy.
* Patients who previously received PD-1 antibody and have experienced toxicities resulting in treatment discontinuation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor-Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab+DC/Myeloma Fusions/GM-CSF: * Nivolumab will be given every two weeks
  * The DC/myeloma fusion vaccine/GM-CSF is administered 4 days per cycle
  Nivolumab: Nivolumab is a monoclonal antibody. Antibodies are part of your immune system; they are a type of protein that protects your body against foreign invaders, called antigens, by grabbing hold of antigens to stop them from invading your system. Nivolumab has been shown to react against cancer cells, including MM cells.
  DC/myeloma fusions/GM-CSF: The DC/MM vaccine is an investigational agent that tries to help the immune system recognize and fight against cancer cells, utilizing unique markers.
Period: Overall Study
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Started (Enrolled and had Tumor and Dendritic Cells Collected) | 5
Initiated Treatment | 2
Completed | 0
Not Completed | 5
Not completed — Lack of Efficacy | 2
Not completed — Progression Prior to Starting Treatment | 3

BASELINE CHARACTERISTICS:
Population: Participants who Initiated Treatment
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 75 [74 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Develop Immunologic Response to Nivolumab and the DC/MM Fusion Vaccine
Description: We planned to evaluate the immunologic response to treatment in blood and bone marrow. Two patients were treated on protocol and both came off due to disease progression early in the course of therapy (one patient during cycle 1 and one patient during cycle 3.) As such, there is insufficient data to perform what had been planned in correlative science studies so no samples were analyzed. This study has been stopped and no further patients are being enrolled and no further samples are being collected. No data has been obtained for any immune analysis; therefore no immune or clinical data will be reported on this trial.
Time Frame: 2 years
Population: Two patients were treated on protocol and both came off due to disease progression early in the course of therapy. Both participants did not achieve a defined clinical response. There is insufficient data to perform what had been planned in correlative science studies or in immune analysis. This study has been stopped and no further patients are being enrolled and no further samples are being collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Number of Patients Who Achieve a Clinical Response (SD, PR, VGPR, CR)
Description: We looked at the two patients who were treated and evaluated their response to treatment.
Time Frame: 2 years
Population: Number of patients who achieved a clinical response
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: We evaluated the number of patients who developed a related adverse event as assessed by the CTCAE version 4.0.
Time Frame: 2 years
Population: Patients who developed treatment-related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Number of Patients Who Are Alive Without Progression at 2 Years
Description: We calculated the number of patients who were alive without progression at 2 years
Time Frame: 2 years
Population: The number of patients who were alive without progression at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of treatment through 30 days after the last dose of treatment up to 6 months. All-Cause Mortality monitored/assessed up to 2 years
Arm/Group | Nivolumab+DC/Myeloma Fusions/GM-CSF
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab+DC/Myeloma Fusions/GM-CSF (N=2)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab+DC/Myeloma Fusions/GM-CSF (N=2)
Alkaline Phosphatase Increase (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Injection Site Reaction (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Muscle Weakness (lower limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, hip (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to withdrawal of funding, this study was halted prematurely. Only two participants were treated and we were unable to analyze the data in any meaningful way due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03782064/Prot_SAP_000.pdf